CLINICAL TRIAL: NCT02634671
Title: Facial Expression Perception by Intensity in Schizophrenia and 22q11.2 Deletion Syndrome: Neural Electrophysiological Evidence by Means of Fast Periodic Visual Stimulation
Brief Title: Perception of Facial Emotions in Schizophrenia and 22q11 Deletion Syndrome
Acronym: FaSchi22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01247- 42
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Facial emotions
MeSH Terms: conditions — Schizophrenia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 22Q11 (Other): 24 patients with 22Q11DS to determine whether the severity of the two disorders' symptoms is correlated with the cerebral response to facial expressions. To answer this question, a set of clinical and neuropsychological tests will be conducted for each patient.
  Interventions: Other: schizophrenia; Other: control group
- SCHIZOPHRENIA (Other): 24 patients with schizophrenia to determine whether the severity of the two disorders' symptoms is correlated with the cerebral response to facial expressions. To answer this question, a set of clinical and neuropsychological tests will be conducted for each patient.
  Interventions: Other: the 22q11 deletion syndrome; Other: control group

INTERVENTIONS:
Other: schizophrenia — The present study aims to identify the mechanisms underlying the deficit in facial emotion recognition reported both in schizophrenia with a control group using an experimental paradigm based on electroencephalography (EEG)
  Arms: 22Q11
Other: the 22q11 deletion syndrome — The present study aims to identify the mechanisms underlying the deficit in facial emotion recognition reported both in the 22q11.2 deletion syndrome with a control group using an experimental paradigm based on electroencephalography (EEG)
  Arms: SCHIZOPHRENIA
Other: control group — The present study aims to identify the mechanisms underlying the deficit in facial emotion recognition reported both in the schizophrenia and 22q11.2 deletion syndrome with a control group using an experimental paradigm based on electroencephalography (EEG)

SUMMARY:
Background:

The present study aims to identify the mechanisms underlying the deficit in facial emotion recognition reported both in schizophrenia and the 22q11.2 deletion syndrome, and thus, reveal a distinction between the two disorders. Indeed, despite the clinical overlap between the two syndromes, some of the symptoms appear to be specific to only one of them. In particular, the disturbance of visual functions is specifically observed in the 22q11.2DS. Hence, the difficulties in facial emotion recognition in schizophrenia and in the 22q11.DS are likely accounted by different cognitive impairments. Investigating which mechanisms are disturbed would allow a specialized support for patients.

Our main hypothesis is that the deficit in facial emotion recognition is more related to visual impairments in the 22q11.2DS than in schizophrenia. This hypothesis will be tested in two groups of patients (22q11.2DS and schizophrenic patients) and a control group (healthy subjects) using an experimental paradigm based on electroencephalography (EEG).

A second aim of this study is to determine whether the severity of the two disorders' symptoms is correlated with the cerebral response to facial expressions. To answer this question, a set of clinical and neuropsychological tests will be conducted for each patient.

DETAILED DESCRIPTION:
Methods:

This study will be conducted using visual steady-state visual evoked potentials (SSVEPs). Visual SSVEPs are periodic neural electrophysiological activities that arise in response to fast periodic visual stimulation (FPVS). They will be recorded in response to the periodic presentation of faces, according to an oddball paradigm. While pictures of faces will appear at a 6 Hz rate, only 1 out of 5 will display an emotion, corresponding to a 1.2 Hz oddball frequency. Different emotions will be tested (happiness, sadness, anger, fear and disgust), displayed with different intensities (20%, 60%, 100%). SSVEPs at 6 Hz will reflect general visual mechanisms (in response to a mixture of low-level (i.e., contrast coding) and high-level (i.e., face detection) processes). Importantly, SSVEPs at 1.2 Hz will index the visual mechanisms specifically involved in facial expression perception and their sensitivity to emotion intensity. Both measures will help determine the underlying brain topographies.

Alongside, clinical and neuropsychological tests will be conducted. While the clinical tests will evaluate the severity of the symptoms, the neuropsychological tests will assess different features such as attention, memory, verbal and visuo-spatial abilities. The patients' scores will be linked with their cerebral activity in response to facial expressions.

Outcomes:

To better understand the impairment of facial emotion recognition in schizophrenia and 22q11.2DS and to improve its care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-50 years old
* No psychiatric conditions or comorbidity
* Agreement from parents if participant is underage
* Patients with schizophrenia: diagnosis assessed with DSM5 criteria
* Patients with 22q11.2 DS: diagnosis assessed by genetic tests (CGH- array or FISH)
* No mental delay (IQ>70 according to the fNART)
* No modification of psychotropic treatment during the month before inclusion

Exclusion Criteria:

* Involvement in a current program of social cognition remediation
* Pregnancy
* Substance use disorder (criteria of DSM-5), except for caffeine and tobacco
* Neurologic disorders (vascular, infectious or neurodegenerative)
* Uncorrected visual deficit
* Guardianship
* Medical drugs with cerebral or psychological effect (e.g, corticosteroids)
* Resistance to antipsychotics
* Electroconvulsive therapy in the previous two months

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10-20 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Steady-state visual evoked potentials (SSVEP) recorded during fast periodic visual stimulation (FPVS). | SSVEPs will be recorded during 20 sequences of emotional faces pictures. As each sequence lasts 80s, the EEG recording will be approximately 30-minutes-long.
  SSVEPs arise in response to the periodic presentation of emotional faces. They are analyzed in the frequency domain. Two types of responses are expected: the general visual response (6 Hz and its harmonics) and the expression-specific response (1.2 Hz and its harmonics). Both responses will be compared across the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: DEMILY CAROLINE, PH, Principal Investigator — Centre régional de dépistage et de prises en charge des troubles psychiatriques d'origine génétique Pôle Ouest LE VINATIER HOSPITAL